CLINICAL TRIAL: NCT04475081
Title: Use of a Live Attenuated Vaccine Repurposed as an Innate Immune-based Preventive Against COVID-19-associated Sepsis/Inflammation
Brief Title: Use of a Live Attenuated Vaccine as an Immune-based Preventive Against COVID-19-associated Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Parsemus Foundation (Unknown)
Responsible Party: Principal Investigator, Paul Fidel, Professor and Associate Dean, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PF-1214
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Sepsis Syndrome
Keywords: MMR vaccine; COVID-19; Sepsis; trained innate immunity; myeloid-derived suppressor cells; inflammation
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; COVID-19; Sepsis; Inflammation | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Intervention Model Description: MMR vaccine vs placebo
Who Masked: Participant
Masking Description: Randomized by study nurse
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MMR vaccination (Experimental): Subjects will be randomized to receive the MMR Vaccine subcutaneously
  Interventions: Biological: MMR vaccine
- Placebo control (Placebo Comparator): Subjects will be randomized to receive sterile saline given subcutaneously
  Interventions: Biological: MMR vaccine

INTERVENTIONS:
Biological: MMR vaccine — Merck MMR-II vaccine

SUMMARY:
The objective of this randomized clinical trial is to test whether administration of live attenuated MMR vaccine (measles mumps rubella; Merck) to eligible adults at highest risk for contracting COVID-19 (healthcare workers, first responders), can induce non-specific trained innate immune leukocytes that can prevent/dampen pathological inflammation and sepsis associated with COVID-19-infection, if exposed.

DETAILED DESCRIPTION:
Clinical Design. Eligible healthcare workers (HCW) or first responders in the greater New Orleans area (n=60) meeting eligibility criteria will be enrolled into a 12 month study by the Louisiana State University Health Sciences Center Clinical & Translational Research Center (LSUHSC CTRC) clinical staff affiliated with the Louisiana Clinical and Translational Research Science (LA CaTS) Center and blindly randomized to receive the live attenuated M-M-R® II vaccine or placebo (sterile saline) via subcutaneous injection in the arm at a baseline visit following informed consent. Subjects will be recruited from local hospitals and EMS stations throughout the greater New Orleans area by distributing recruitment flyers at the local facilities. The flyers will have contact information for HCWs and EMS first responders to call for more information or to schedule an appointment. Additionally, subjects may be referred to the study by other HCWs or first responders aware of study activities. Subject consenting, interviewing, vaccine administration and biospecimen collection will be performed by the CTRC staff, under full Personal Protective Equipment (PPE) protection. Following informed consent, subjects will be asked to complete the Baseline Demographic & History Questionnaire disclosing their demographic information, employment, medication, vaccination, and medical history. Specifically, the medical history will place emphasis on the presence of diabetes, hypertension, heart disease, and their treatments/medications. Subjects will then have their height, weight, body mass index (BMI), vital signs, and pulse oximetry measured. Subjects will also have their body composition and fat percentage measured using the BOD POD Body Composition Tracking System. Female subjects of childbearing potential will be given a urine-based pregnancy test. Approximately 10cc of blood will be collected along with a nasopharyngeal swab for baseline laboratory analyses (serology, RNA, flow cytometry). When available, a finger prick blood sample will be obtained in addition to the other biospecimens for COVID-19 serological analysis. Those subjects that satisfy the inclusion and exclusion criteria (Eligibility Criteria) will be blindly randomized to receive the live attenuated M-M-R® II vaccine or placebo (sterile saline) via subcutaneous injection. Repeat biosampling will occur on days 30, 60, and at 12 months post-vaccination. At each follow-up, anthropometric measurements, vital signs measurement, and symptom assessment for the presence of symptoms related to COVID-19 infection (fever, headache, myalgia, cough, loss of taste or smell, breathing problems), general well-being (i.e., pain, dental concerns, sleep patterns, general stress level, fatigue), and any changes in medications, medical status, and employment will be collected utilizing the Follow-up Symptom & History Questionnaire. Telephone follow-up calls utilizing the Follow-up Symptom Assessment & History Questionnaire will be made on a monthly basis between the 60-day follow-up visit and the 12-month endpoint visit. Should a subject develop symptoms potentially associated with COVID-19 infection at any point during the 12-month study period, that subject will be seen in the clinic by the Infectious Disease (ID) Co-investigator, and a repeat collection of blood and nasopharyngeal biospecimens will be performed for analysis, and the subject will be asked to complete the Follow-up Symptom & History Questionnaire and get another body composition analysis via BOD POD. Subjects will be asked to report the development of any potential COVID-19 infection-related symptoms or positive COVID-19 infection testing outside of the study, as well as any symptoms potentially related to MMR vaccination. Should a subject become admitted to the hospital related to COVID-19 infection, in-patient information will be obtained via the electronic medical record (EMR) when available.

Primary outcome measures will be peripheral blood monocytic MDSCs (M-MDSC) and/or granulocytic MDSCs (G-MDSC) determined by flow cytometry from whole blood samples. Specifically, documented increases in the MDSCs per subject from baseline through 30-60 days post-vaccination is expected in the MMR group compared to placebo group. Measles antibody are also expected to increase in the MMR group and will serve as a control for the MMR vaccination. Stationary levels of MDSCs and measles antibodies are expected in the MMR group over the 12-month period.

The investigators will perform the COVID-19 RNA testing at baseline, 30, and 60 days post-vaccination, and at any point over the 12-month period that symptoms arise. All patients that are COVID-19+ at baseline or become COVID-19+ through the study will be included for secondary outcome analyses. The Secondary outcome measures will be COVID-19 antibodies (seropositive) as evidence of infection, sepsis/lung inflammation, ICU/ventilator usage, in-patient health related co-morbidities and self-reporting mental status (such as general fatigue/stress level) over the 12-month period post-vaccination. In-patient information will be obtained through the EMR when available. Out-patient information will be obtained via self-reporting utilizing the Follow-up Symptom & History Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* Employed as a HCW (hospital, outpatient clinic, private office or 1st responder (EMS) in the greater New Orleans region
* Able to provide a signed and dated informed consent
* Able to provide pre-randomized blood specimen

Exclusion Criteria:

* Any known MMR vaccine contraindication
* Fever
* Weakened resistance toward infections due to a disease in/of the immune system
* Individuals receiving medical treatment that affects the immune response or other immunosuppressive therapy in the last year (see excluded medications).
* Individuals with a congenital cellular immunodeficiency
* Individuals with a malignancy involving bone marrow or lymphoid systems
* Individuals with any serious underlying illness (such as malignancy). People with cardiovascular disease, hypertension, diabetes, and/or chronic respiratory disease are eligible if not immunocompromised (at the discretion of the ID Co-investigator)
* Individuals with known or suspected HIV infection, even if asymptomatic or has normal immune function. (Due to the risk of disseminated MMR infection)
* Individuals with an active skin disease such as eczema, dermatitis or psoriasis at or near the site of vaccination. A different site can be chosen if necessary
* Pregnant or women who think they may test positive for pregnancy in this next month following MMR vaccine administration.
* Individuals who have received a MMR or another live vaccine (i.e., Zostavax, nasal flu vaccine) within the last year
* Individuals with known anaphylactic reaction to any of the ingredients present in the MMR vaccine
* Individuals previously testing positive for SARS-CoV-2 or documented seropositive for SARS-CoV-2 antibodies prior to enrollment in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Fidel, PhD, Principal Investigator — Louisiana State University Health Sciences Center - New Orleans
Locations (1):
- Clinical and Translational Research Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified participant data to other researchers at their request and with justification. Primary and secondary outcome measures will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: If fully justified for additional research purposes

REFERENCES:
- [Background] Fidel PL Jr, Noverr MC. Could an Unrelated Live Attenuated Vaccine Serve as a Preventive Measure To Dampen Septic Inflammation Associated with COVID-19 Infection? mBio. 2020 Jun 19;11(3):e00907-20. doi: 10.1128/mBio.00907-20. PMID 32561657
- [Derived] Noverr MC, Yano J, Hagensee ME, Lin HY, Meyaski MC, Meyaski E, Cameron J, Shellito J, Trauth A, Fidel PL Jr. Effect of MMR Vaccination to Mitigate Severe Sequelae Associated With COVID-19: Challenges and Lessons Learned. Med Res Arch. 2023 Feb;11(2):3598. doi: 10.18103/mra.v11i2.3598. PMID 37153751

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MMR Vaccination | Placebo Control
Started | 25 | 25
Completed | 19 | 15
Not Completed | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MMR Vaccination | Placebo Control | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 10 | 27
  >=65 years | 2 | 5 | 7
Age, Continuous [Median (Full Range); unit: years] | 51 [27 to 75] | 55 [25 to 81] | 52 [25 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 17 | 14 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 16 | 12 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 15 | 34

OUTCOME MEASURES:

1. Primary Outcome: Induction of MDSCs
Description: peripheral blood monocytic MDSCs (M-MDSC) and/or granulocytic MDSCs (G-MDSC) determined by flow cytometry from whole blood samples as percentage/fold change over baseline
Time Frame: 30 days post vaccination
Population: Myeloid-derived suppressor cells in blood
Measure: Mean (Standard Deviation); unit: fold change compared to baseline
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
fold change compared to baseline | 0.19 (0.19) | 0.11 (0.17)

2. Primary Outcome: Induction of MDSCs
Description: as for outcome 1
Time Frame: 60 days post vaccination
Population: Myeloid-derived suppressor cells in blood
Measure: Mean (Standard Deviation); unit: fold change compared to baseline
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
fold change compared to baseline | 0.19 (0.19) | 0.25 (0.25)

3. Primary Outcome: Induction of MDSCs
Description: as for outcome 1
Time Frame: 12 months post vaccination
Population: Myeloid-derived suppressor cells
Measure: Mean (Standard Deviation); unit: fold change compared to baseline
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
fold change compared to baseline | 0.09 (0.08) | 0.09 (0.12)

4. Secondary Outcome: COVID-19 Infection Positive
Description: COVID-19 antibodies (seropositive) or COVID-19 RNA+ as evidence of infection
Time Frame: 30 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

5. Secondary Outcome: COVID-19 Infection Positive
Description: COVID-19 antibodies (seropositive) or COVID-19 RNA+ as evidence of infection
Time Frame: 60 days post-vaccination
Population: positive test for COVID-19 - antibodies or PCR
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

6. Secondary Outcome: COVID-19 Infection Positive
Description: COVID-19 antibodies (seropositive) or COVID-19 RNA+ as evidence of infection
Time Frame: 12 months post-vaccination
Population: positive test for COVID-19 - antibodies or PCR
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 1 | 0

7. Secondary Outcome: Health Questionnaire
Description: Sepsis/lung inflammation, ICU/ventilator usage, in-patient health related co-morbidities and self-reporting mental status (such as general fatigue/stress level)
Time Frame: 14 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

8. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 30 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

9. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 60 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

10. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 3 months post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

11. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 4 months post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

12. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 5 months post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

13. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 6 months post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

14. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 7 months post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

15. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 8 months post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

16. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 9 months post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

17. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 10 months post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

18. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 11 months post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

19. Secondary Outcome: Health Questionnaire
Description: as for outcome 7
Time Frame: 12 months post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | MMR Vaccination | Placebo Control
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 72 h post-vaccination for any allergic responses. After 72 h allergic responses would not be evident. Any other monitoring for adverse events and conditions were monitored monthly through a 12-month enrollment period in the study
Description: allergic reactions to the vaccine were monitored by calls by nursing staff or reported back to nursing staff over a 72 h period post-vaccination. Any other adverse events, treatment or non-treatment, were monitored by the nursing staff via monthly phone calls. Adverse events could have been any type of sickness, including COVID. Any adverse events would be recorded and documented, but only those related to COVID would be part of the results obtained and used in the analyses.
Arm/Group | MMR Vaccination | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/15
Other Adverse Events (participants affected / at risk) | 0/19 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMR Vaccination (N=19) | Placebo Control (N=15)
allergy (Immune system disorders) | 1 (1) | 0 (0) — Allergic reaction to the MMR vaccine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT04475081/Prot_SAP_002.pdf
  • Informed Consent Form (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT04475081/ICF_003.pdf